CLINICAL TRIAL: NCT02287922
Title: A Phase IIb Multicenter, Randomized, Double-blind Study of ALX-0061 Administered Subcutaneously as Monotherapy, in Subjects With Moderate to Severe Rheumatoid Arthritis Who Are Intolerant to Methotrexate or for Whom Continued Methotrexate Treatment is Inappropriate
Brief Title: A Phase IIb Study for ALX-0061 Monotherapy in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALX0061-C202; 2014-003012-36 (EudraCT Number)
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ALX-0061; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ALX-0061 150 mg q4w (Experimental): ALX-0061 150 mg every 4 weeks from baseline through Week 12 + placebo every 2 weeks from baseline through Week 12. The last injection with study drug was administered at the Week 10 visit.
  Interventions: Biological: ALX-0061; Biological: Placebo
- ALX-0061 150 mg q2w (Experimental): ALX-0061 150 mg every 2 weeks from baseline through Week 12 + placebo every 2 weeks from baseline through Week 12. The last injection with study drug was administered at the Week 10 visit.
  Interventions: Biological: ALX-0061; Biological: Placebo
- ALX-0061 225 mg q2w (Experimental): ALX-0061 225 mg every 2 weeks from baseline through Week 12. The last injection with study drug was administered at the Week 10 visit.
  Interventions: Biological: ALX-0061
- TCZ 162 mg q1w or q2w (Active Comparator): Open-label TCZ. Injections were to be performed q1w or q2w depending on the approved label per region (last injection was administered at Week 10 or Week 11, depending on the dose regimen).
  Interventions: Biological: Tocilizumab

INTERVENTIONS:
Biological: ALX-0061
  Arms: ALX-0061 150 mg q2w; ALX-0061 150 mg q4w; ALX-0061 225 mg q2w
Biological: Placebo
  Arms: ALX-0061 150 mg q2w; ALX-0061 150 mg q4w
Biological: Tocilizumab
  Arms: TCZ 162 mg q1w or q2w

SUMMARY:
The primary objective of this study is:

- To assess the efficacy and safety of dose regimens of ALX-0061 monotherapy administered subcutaneously (s.c.) to subjects with active rheumatoid arthritis (RA).

The secondary objectives of this study are:

* To assess the effects of ALX-0061 on quality of life, the pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of ALX-0061 and to explore potential dose regimens for ALX-0061 monotherapy, based on safety and efficacy, for further clinical development.
* To obtain parallel descriptive information concerning the efficacy and safety of tocilizumab (TCZ) s.c. in the same clinical trial RA population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA (according to the 2010 EULAR/American College of Rheumatology (ACR) classification criteria) for at least 6 months prior to screening, and ACR functional class I-III.
* Received previous or current treatment with methotrexate (MTX), and is considered intolerant to MTX, or for whom continued treatment with MTX is inappropriate or has contraindications for MTX use.
* Subjects must not have received MTX for at least 4 weeks before first administration of the study drug.
* Have active RA with at least 6 swollen and 6 tender joints(66/68 joint count) at the time of screening and baseline
* Others as defined in the protocol

Exclusion Criteria:

* Have been treated with DMARDs (Disease Modifying Antirheumatic Drugs)/systemic immunosuppressive drugs during the 4 weeks, or 12 weeks for hydroxychloroquine, chloroquine, or leflunomide (except when an adequate wash-out procedure for leflunomide was completed), prior to first administration of study drug.
* Have received approved or investigational biological or targeted synthetic DMARD therapies for RA (including tumor necrosis factor alpha-inhibitors, abatacept, rituximab, or Janus kinase [JAK]-inhibitors) less than 6 months prior to screening.
* Have a history of toxicity, non-tolerance, primary non-response or inadequate response to a biological therapy, or targeted synthetic DMARDs (including JAK inhibitors), for RA.
* Have received prior therapy blocking the interleukin-6 (IL-6) pathway, at any time.
* Others as defined in the protocol.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Ablynx, a Sanofi company
Locations (80):
- United States (17):
  - Investigator Site, Birmingham, Alabama
  - Investigator Site, Hemet, California
  - Investigator Site, La Palma, California
  - Investigator site, Los Angeles, California
  - Investigator Site, Los Angeles, California
  - Investigator site, Ventura, California
  - Investigator site, Hialeah, Florida
  - Investigator Site, Homestead, Florida
  - Investigator Site, Orlando, Florida
  - Investigator Site, Stockbridge, Georgia
  - Investigator site, Overland Park, Kansas
  - Investigator Site, Worcester, Massachusetts
  - Investigator Site, Albuquerque, New Mexico
  - Investigator Site, New York, New York
  - Investigator Site, Charleston, South Carolina
  - Investigator Site, Memphis, Tennessee
  - Investigator Site, Mesquite, Texas
- Belgium (3):
  - Investigator Site, Brussels
  - Investigator Site, Ghent
  - Investigator Site, Liège
- Bulgaria (7):
  - Investigator Site, Burgas
  - Investigator Site, Pleven
  - Investigator Site 1, Plovdiv
  - Investigator Site 2, Plovdiv
  - Investigator Site 1, Rousse
  - Investigator Site 2, Rousse
  - Investigator Site, Sofia
- Czechia (6):
  - Investigator Site, Brno
  - Investigator Site, Olomouc
  - Investigator Site, Ostrava
  - Investigator Site 1, Prague
  - Investigator Site 2, Prague
  - Investigator Site, Zlín
- Georgia (3):
  - Investigator Site, Tbilisi
  - Investigator Site 1, Tbilisi
  - Investigator Site 2, Tbilisi
- Germany (3):
  - Investigator Site, Berlin
  - Investigator Site, Frankfurt
  - Investigator Site, Hamburg
- Hungary (8):
  - Investigator Site, Baja
  - Investigator Site, Budapest
  - Investigator Site, Esztergom
  - Investigator site, Gyula
  - Investigator Site, Székesfehérvar
  - Investigator Site, Szikszó
  - Investigator Site, Szombathely
  - Investigator Site, Veszprém
- Mexico (7):
  - Investigator Site, Culiacán
  - Investigator Site, León
  - Investigator Site 1, Mexico City
  - Investigator Site 2, Mexico City
  - Investigator Site, Mexico City
  - Investigator Site 1, Monterrey
  - Investigator Site 2, Monterrey
- Investigator Site, Chisinau, Moldova
- North Macedonia (2):
  - Investigator Site 1, Skopje
  - Investigator Site 2, Skopje
- Poland (10):
  - Investigator Site, Bydgoszcz
  - Investigator Site 2, Elblag
  - Investigator Site, Elblag
  - Investigator Site, Gdynia
  - Investigator Site, Grodzisk Mazowiecki
  - Investigator Site, Lublin
  - Investigator SIte, Poznan
  - Investigator Site, Sochaczew
  - Investigator Site, Torun
  - Investigator Site, Warsaw
- Romania (3):
  - Investigator Site, Bucharest
  - Investigator Site, Oradea
  - Investigator Site, Timișoara
- Serbia (4):
  - Investigator Site 1, Belgrade
  - Investigator Site 2, Belgrade
  - Investigator Site 3, Belgrade
  - Investigator Site, Niška Banja
- Spain (6):
  - Investigator Site, Córdoba
  - Investigator Site, Madrid
  - Investigator Site, Santander
  - Investigator Site 2, Santander
  - Investigator Site 1, Santiago de Compostela
  - Investigator Site 2, Santiago de Compostela

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 251 subjects were recruited at 58 sites located in Europe (42 sites; 199 subjects), Latin America (6 sites; 36 subjects) and North America (10 sites; 16 subjects). Consent was obtained from the first subject on 18 Mar 2015; the last subject completed the final visit in on 19 Jul 2016.
Pre-assignment Details: Of the 599 subjects screened, 348 were screen failures and 251 subjects were randomly assigned to treatment (Intent-to-treat population). All subjects enrolled received study treatment and were included in the safety population. All subjects who received at least one dose of ALX-0061 were included in the pharmacokinetic (PK) population.
Groups:
- ALX-0061 150 mg q4w: ALX-0061 150 mg every 4 weeks from baseline through Week 12 + placebo every 2 weeks from baseline through Week 12. The last injection with study drug was administered at the Week 10 visit.
  ALX-0061
  Placebo
- ALX-0061 150 mg q2w: ALX-0061 150 mg every 2 weeks from baseline through Week 12 + placebo every 2 weeks from baseline through Week 12. The last injection with study drug was administered at the Week 10 visit.
  ALX-0061
  Placebo
- ALX-0061 225 mg q2w: ALX-0061 225 mg every 2 weeks from baseline through Week 12. The last injection with study drug was administered at the Week 10 visit.
  ALX-0061
- TCZ 162 mg q1w or q2w: Open-label tocilizumab (TCZ). Injections were to be performed q1w or q2w depending on the approved label per region (last injection was administered at Week 10 or Week 11, depending on the dose regimen).
  Tocilizumab
Period: Overall Study
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Started | 62 | 62 | 63 | 64
Completed | 59 | 60 | 56 | 57
Not Completed | 3 | 2 | 7 | 7
Not completed — Adverse Event | 1 | 1 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Sponsor's decision | 0 | 0 | 0 | 1
Not completed — Other | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- TCZ 162 mg q1w or q2w: Open-label TCZ. Injections were to be performed q1w or q2w depending on the approved label per region (last injection was administered at Week 10 or Week 11, depending on the dose regimen).
  Tocilizumab
- Total: Total of all reporting groups
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w | Total
Number analyzed (Participants) | 62 | 62 | 63 | 64 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 1
  Between 18 and 65 years | 50 | 53 | 56 | 58 | 217
  >=65 years | 12 | 8 | 7 | 6 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (12.25) | 51.2 (12.05) | 51.3 (11.81) | 50.0 (12.26) | 51.4 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 53 | 54 | 56 | 212
  Male | 13 | 9 | 9 | 8 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects With American College of Rheumatology 20 (ACR20) at Week 12
Description: ACR 20 response is defined as:
  * 20% improvement in tender joint count (TJC; 68 joints) relative to Week 0 AND
  * 20% improvement in swollen joint count (SJC; 66 joints) relative to Week 0 AND
  * 20% improvement in 3 of the following 5 areas relative to Week 0:
    * Subject's Assessment of Pain (100 mm - visual analogue scale [VAS])
    * Subject's Global Assessment of Disease Activity (VASPA)
    * Physician's Global Assessment of Disease Activity (VASPHA)
    * Subject's assessment of physical function as measured by Health Assessment Questionnaire-Disability Index (HAQ-DI)
    * C-reactive protein (CRP) level
  The primary endpoint was analyzed using non-responder imputation (NRI), i.e., subjects with missing ACR20 response at Week 12 were treated as non-responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 45 | 48 | 51 | 50

2. Secondary Outcome: Number and Percentage of Subjects With ACR50 and ACR70 Response at Week 12
Description: ACR50/70 response is defined as:
  * 50/70% improvement in TJC (68 joints) relative to Week 0 AND
  * 50/70% improvement in SJC (66 joints) relative to Week 0 AND
  * 50/70% improvement in 3 of the following 5 areas relative to Week 0:
    * Subject's Assessment of Pain (100 mm - VAS)
    * Subject's Global Assessment of Disease Activity (VASPA)
    * Physician's Global Assessment of Disease Activity (VASPHA)
    * Subject's assessment of physical function as measured by HAQ-DI
    * CRP level
  This endpoint was analyzed using NRI, i.e., subjects with missing response at Week 12 were treated as non-responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants
  ACR50 | 27 | 23 | 31 | 29
  ACR70 | 10 | 15 | 13 | 15

3. Secondary Outcome: Number and Percentage of Subjects With Low Disease Activity (LDA) Using Disease Activity Score Using 28 Joint Counts (DAS28) Using C-reactive Protein (CRP) at Week 12
Description: DAS28(CRP) = (0.56 × √TJC28) + (0.28 × √SJC28) + (0.36 × ln[CRP+1]) + (0.014 × VASPA) + 0.96
  Low disease activity = 2.6 ≤ DAS28 ≤ 3.2
  Subjects with low disease activity includes subjects who are in remission. This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non-responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 26 | 35 | 38 | 28

4. Secondary Outcome: Number and Percentage of Subjects With LDA Using DAS28 Using Erythrocyte Sedimentation Rate (ESR) at Week 12
Description: DAS28(ESR) = (0.56 × √TJC28) + (0.28 × √SJC28) + (0.70 × ln[ESR]) +(0.014 × VASPA)
  Low disease activity = 2.6 ≤ DAS28 ≤ 3.2
  Subjects with low disease activity includes subjects who are in remission. This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non-responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 26 | 32 | 34 | 20

5. Secondary Outcome: Number and Percentage of Subjects With LDA Using Simplified Disease Activity Index (SDAI) at Week 12
Description: SDAI = TJC28 + SJC28 + VASPA + VASPHA + CRP (mg/dL)
  Low disease activity: 3.3 < SDAI ≤ 11.0
  Subjects with low disease activity includes subjects who are in remission. This endpoint was analyzed using non-responder imputation (NRI), i.e., subjects with missing response at the concerned visit were treated as non-responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 23 | 27 | 33 | 22

6. Secondary Outcome: Number and Percentage of Subjects With LDA Using Clinical Disease Activity Index (CDAI) at Week 12
Description: CDAI = TJC28 + SJC28 + VASPA + VASPHA
  Low disease activity: 2.8 < CDAI ≤ 10
  Subjects with low disease activity includes subjects who are in remission. This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non-responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 23 | 21 | 32 | 21

7. Secondary Outcome: Number and Percentage of Subjects With European League Against Rheumatism (EULAR) (CRP) Good Response at Week 12
Description: EULAR good response is defined as an improvement of >1.2 in DAS28 (CRP) relative to baseline.
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non-responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 25 | 34 | 38 | 28

8. Secondary Outcome: Number and Percentage of Subjects in Remission Using DAS28 (ESR) at Week 12
Description: DAS28(ESR) = (0.56 × √TJC28) + (0.28 × √SJC28) + (0.70 × ln[ESR]) +(0.014 × VASPA)
  Remission = DAS28(ESR) < 2.6
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non-responders.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 21 | 13 | 25 | 16

9. Secondary Outcome: Number and Percentage of Subjects in Remission Using SDAI at Week 12
Description: SDAI = TJC28 + SJC28 + VASPA + VASPHA + CRP (mg/dL)
  Remission: SDAI ≤ 3.3
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non-responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 5 | 3 | 5 | 7

10. Secondary Outcome: Number and Percentage of Subjects in Remission Using CDAI at Week 12
Description: CDAI = TJC28 + SJC28 + VASPA + VASPHA
  Remission: CDAI ≤ 2.8
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non-responders.
Time Frame: Week 12
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 6 | 3 | 4 | 6

11. Secondary Outcome: Number and Percentage of Subjects in Remission Using Boolean Defined Remission Criteria at Week 12
Description: Boolean remission: tender joint count (TJC)28 ≤ 1 and swollen joint count (SJC)28 ≤ 1 and VASPA (cm) ≤ 1 and CRP (mg/dL) ≤ 1
  This endpoint was analyzed using NRI, i.e., subjects with missing response at the concerned visit were treated as non-responders.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 2 | 3 | 4 | 4

12. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 12
Description: The HAQ-DI is a 20-question instrument which assesses the degree of difficulty the subject had in accomplishing tasks in 8 functional areas over the previous week. The 8 areas are: dressing and grooming, hygiene, arising, reach, eating, grip, walking, common daily activities. Within each area, subjects report the amount of difficulty they have in performing the specific items. There are 4 response options ranging from: 0 = No Difficulty, 1 = With Some Difficulty, 2 = With Much Difficulty, 3 = Unable to Do. The 8 areas are each given a single score equal to the maximum value of their component activities (0, 1, 2, or 3). The sum of the area scores is then divided by the number of areas answered to obtain the final HAQ score (rounded to the nearest value evenly divisible by 0.125). The final HAQ-DI score ranges from 0 to 3. A high score means a high degree of disability (=worse outcome).
  Missing values were imputed with the last non-missing observation.
Time Frame: From baseline until Week 12
Population: Intent-to-treat population, number of participants with data available
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 61 | 60 | 59 | 64
score on a scale | -0.541 (0.0809) | -0.746 (0.0935) | -0.817 (0.0802) | -0.689 (0.0811)

13. Secondary Outcome: Change From Baseline in Physical and Mental Component Scores of Short Form Health Survey (SF-36) at Week 12
Description: The Short Form (36) Health Survey (SF-36) consists of 36 items that can be summarized into 8 domains: physical functioning, role limitations due to physical health problems (role-physical), bodily pain, general health, vitality, social functioning, role limitations due to emotional problems (role-emotional), and mental health. Two summary measures, the physical component summary and the mental component summary, can be derived based on these domain scores. Each score is directly transformed into a 0-100 score on the assumption that each question carries equal weight. Low score indicates greater disability.
Time Frame: From baseline until week 12
Population: Intent-to-treat population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
score on a scale
  physical component: number analyzed (Participants) | 58 | 60 | 56 | 54
  physical component | 7.808 (0.8533) | 7.979 (1.1895) | 8.861 (1.0818) | 7.611 (0.9562)
  mental component: number analyzed (Participants) | 58 | 60 | 56 | 55
  mental component | 5.49 (1.221) | 8.836 (1.5243) | 8.913 (1.3903) | 6.156 (1.3192)

14. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Subscale at Week 12
Description: The FACIT Measurement System is a collection of health-related quality of life questionnaires that assess multidimensional health status in people with various chronic illnesses. The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued). To score the FACIT-fatigue, all items are summed to create a single fatigue score with a range from 0 to 52. Items are reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue.
Time Frame: From baseline until Week 12
Population: Intent-to-treat population, number of subjects with data available
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 58 | 60 | 56 | 57
score on a scale | 7.832 (1.3438) | 11.41 (1.53) | 12.996 (1.3702) | 8.971 (1.4461)

15. Secondary Outcome: Pharmacodynamics: Concentrations of Soluble Interleukin-6 Receptor (sIL-6R)
Description: Values below the limit of quantification are imputed with the lower limit of quantification (LLOQ).
Time Frame: From baseline until Week 12
Population: Safety population
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
ng/mL
  Baseline | 33.0 (4.65) | 42.3 (8.71) | 30.9 (3.72) | 31.0 (2.54)
  Week 12: number analyzed (Participants) | 58 | 59 | 56 | 56
  Week 12 | 376 (21.6) | 460 (19.9) | 459 (18.8) | 269 (11.1)

16. Secondary Outcome: Pharmacokinetics: ALX-0061 Concentration in Serum at Week 12
Time Frame: From baseline until Week 12
Population: PK Population, participants with data available
Measure: Geometric Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w
Number analyzed (Participants) | 54 | 55 | 52
micrograms/milliliter | 1.4 (3.61) | 18.4 (2.95) | 27.9 (2.53)

17. Secondary Outcome: Number and Percentage of Subjects With Development of a Treatment-emergent Antidrug Antibody Response
Time Frame: From first study drug intake up to and including follow-up (FU), i.e., maximum of 22 weeks (10 weeks of treatment + 12 weeks of FU)
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- ALX-0061 Total: This group includes all participants who received at least one dose of ALX-0061
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | ALX-0061 Total
Number analyzed (Participants) | 62 | 62 | 63 | 187
Participants | 7 | 25 | 26 | 58

18. Secondary Outcome: Number and Percentage of Subjects With Treatment-emergent Adverse Event by Severity
Time Frame: From baseline until Week 12
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants
  Mild | 22 | 18 | 21 | 19
  Moderate | 12 | 13 | 9 | 10
  Severe | 0 | 2 | 1 | 2

19. Secondary Outcome: Number of Treatment-emergent Adverse Event by Severity
Time Frame: From baseline until Week 12
Population: Safety population
Measure: Number; unit: Treatment-emergent adverse events
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Treatment-emergent adverse events
  Mild | 46 | 75 | 84 | 47
  Moderate | 18 | 22 | 15 | 15
  Severe | 0 | 2 | 3 | 2

20. Secondary Outcome: Number and Percentage of Subjects With a Treatment-related Treatment-emergent Adverse Event
Description: treatment related = considered at least possibly related to study drug by the Investigator
Time Frame: From baseline until Week 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
Participants | 21 | 20 | 21 | 20

21. Secondary Outcome: Number of Treatment-related Treatment-emergent Adverse Event
Description: treatment related = considered at least possibly related to study drug by the Investigator
Time Frame: From baseline until Week 12
Population: Safety Population
Measure: Number; unit: treatment-emergent adverse events
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
Number analyzed (Participants) | 62 | 62 | 63 | 64
treatment-emergent adverse events | 46 | 53 | 64 | 32

ADVERSE EVENTS:
Time Frame: From first study drug intake up to and including follow-up, i.e., maximum of 22 weeks when assigned to the ALX-0061 or TCZ q2w treatment groups (10 weeks of treatment + 12 weeks of follow-up), or 23 weeks when assigned to the TCZ q1w treatment group (11 weeks of treatment + 12 weeks of follow-up)
Arm/Group | ALX-0061 150 mg q4w | ALX-0061 150 mg q2w | ALX-0061 225 mg q2w | TCZ 162 mg q1w or q2w
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/62 | 0/62 | 2/63 | 2/64
Other Adverse Events (participants affected / at risk) | 15/62 | 20/62 | 17/63 | 12/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALX-0061 150 mg q4w (N=62) | ALX-0061 150 mg q2w (N=62) | ALX-0061 225 mg q2w (N=63) | TCZ 162 mg q1w or q2w (N=64)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail bed infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALX-0061 150 mg q4w (N=62) | ALX-0061 150 mg q2w (N=62) | ALX-0061 225 mg q2w (N=63) | TCZ 162 mg q1w or q2w (N=64)
Alanine aminotransferase increased (Infections and infestations) | 1 (1) | 0 (0) | 4 (5) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 1 (1) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 3 (3) | 0 (0) | 5 (5)
Injection site erythema (General disorders) | 4 (7) | 7 (10) | 5 (20) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of any results from this study will be according to the principles of the Declaration of Helsinki and will require prior review and written agreement of the Sponsor.

DOCUMENTS (1):
  • Study Protocol (2015-07-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT02287922/Prot_000.pdf